CLINICAL TRIAL: NCT06267495
Title: Epithelium-on Accelerated Corneal Cross-linking Versus Observation of Fellow Eyes of Young Patients With Unilateral Clinically Evident Keratoconus
Brief Title: Epithelium-on Cross-linking Versus Observation of Fellow Eyes of Patients With Unilateral Clinically Evident Keratoconus
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdel-Radi, Principal Investigator, Assiut University
Other Study IDs: EOCXLFE
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Keratoconus
Keywords: Keratoconus; Corneal cross-linking; Epithelium-on CXL
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Epithelium-on corneal cross-linking group: Patients in this group underwent epithelium-on accelerated corneal cross-linking (epi-on CXL) for the eye with no clinical signs of keratoconus.
  Interventions: Procedure: Epithelium-on corneal cross-linking (epi-on CXL)
- Follow-up group: Patients in this group were planned to have regular follow-up visits, without intervention, for the eye with no clinical signs of keratoconus.

INTERVENTIONS:
Procedure: Epithelium-on corneal cross-linking (epi-on CXL) — In epithelium-on corneal cross-linking (epi-on CXL), the cornea is soaked with riboflavin for 10 minutes (Paracel® for 4 minutes and VibeX-xtra® for 6 minutes) . Thereafter, the cornea is subjected to ultraviolet A at a wavelength of 370 nm to give a total dose of 5.4 J/cm² through 10 milliwatt mW/cm² for 9 minutes.
  Groups: Epithelium-on corneal cross-linking group

SUMMARY:
Keratoconus (KC) is a bilateral asymmetric progressive corneal degenerative disease. The management of young patients, diagnosed with clinically evident KC in one eye and with no clinical signs of KC in the other eye, represents a real challenge for many ophthalmologists.

The aim of the current study is to investigate the effectiveness and safety of epithelium-on accelerated CXL to stabilize the eye with no clinical signs of KC, in young patients with unilateral clinically evident KC, compared with standard care and follow-up only.

DETAILED DESCRIPTION:
Keratoconus (KC) is a bilateral asymmetric progressive corneal degenerative disease associated with corneal thinning and protrusion with resultant irregular astigmatism and visual loss.

Although several studies showed that epithelium-off corneal cross-linking (epi-off CXL) is more effective in preventing KC progression compared with epithelium-on corneal cross-linking (epi-on CXL), the removal of corneal epithelium in epi-off CXL might be associated with a number of serious complications such as persistent epithelial defects and sight-threatening infectious keratitis. Additionally, recent systematic reviews and meta-analysis concluded that epi-on CXL is as effective as epi-off CXL in terms of visual and topographic stability of keratoconus, but has the advantage of being much safer avoiding the complications of epithelial removal.

The management of the better eye, of young patients with unilateral clinically evident KC, is controversial. Some ophthalmologists prefer to cross-link the better eye, while others prefer to conservatively follow it up, in order to avoid complications of epithelial removal in epi-off CXL.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 12 to 30 years presented with forme fruste (FFKC) or subclinical KC, based on the following criteria:

1. Normal slit lamp examination
2. Normal topography in FFKC and suspicious topography in subclinical KC with asymmetric bow-tie or inferior steeping (inferior-superior value less than 1.40 D in the anterior sagittal curvature map in pentacam)
3. Clinical and topographic features of KC in the other eye.

Exclusion Criteria:

1. Corrected distance visual acuity (CDVA) worse than 0.1 logMAR
2. Corneal thickness at the thinnest location less than 400 μm
3. Severe ocular allergy (active catarrhal keratoconjunctivitis)
4. Other corneal or ocular diseases
5. Systemic diseases such as diabetes mellitus and autoimmune diseases

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This retrospective comparative study was conducted at a refractive and corneal surgery center in Assiut (Private practice). The study included young patients who were diagnosed with forme fruste or subclinical keratoconus.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Steep keratometry value | 24 months
  The steep keratometry is measured using pentacam. A higher value means a worse outcome.
Maximum keratometry value | 24 months
  The maximum keratometry is measured using pentacam. A higher value means a worse outcome.

SECONDARY OUTCOMES:
Corrected distance visual acuity | 24 months
  Corrected distance visual acuity (CDVA) is measured with Snellen's acuity chart and converted to logarithm of the minimum angle of resolution (logMAR) notation.
  The higher the logMAR CDVA, the worse the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Abdel-Radi, MD, Principal Investigator — Assiut University
Locations (1):
- Tiba Eye Center, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koh S, Inoue R, Maeda N, Kabata D, Shintani A, Jhanji V, Klyce SD, Maruyama K, Nishida K. Long-term Chronological Changes in Very Asymmetric Keratoconus. Cornea. 2019 May;38(5):605-611. doi: 10.1097/ICO.0000000000001890. PMID 30702472
- [Background] Henriquez MA, Hadid M, Izquierdo L Jr. A Systematic Review of Subclinical Keratoconus and Forme Fruste Keratoconus. J Refract Surg. 2020 Apr 1;36(4):270-279. doi: 10.3928/1081597X-20200212-03. PMID 32267959